CLINICAL TRIAL: NCT02180633
Title: Unveiling Preclinical Idiopathic Macular Hole Formation
Acronym: IMH_2012
Status: Completed | Type: Observational
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Rui Bernardes, Prof., University of Coimbra
Other Study IDs: BBB-BMD/2739/2012
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Idiopathic Macular Hole
Keywords: Idiopathic Macular Hole

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Fellow Eyes: Patients that suffer from unilateral idiopathic macular hole, and whose fellow eyes don't show any sign of retinal pathology.
  Interventions: Other: Optical Coherence Tomography Scan
- Controls: Healthy subjects age-matched to the other group, with no visible retinal pathologies.
  Interventions: Other: Optical Coherence Tomography Scan

INTERVENTIONS:
Other: Optical Coherence Tomography Scan — As an observational study, the only interventive action taken is the acquisition of a non-invasive volumetric image of the retina via optical coherence tomography (OCT).

SUMMARY:
A macular hole is a rupture in the macula. In terms of pathogenesis, as much as 80% are idiopathic (Idiopathic Macular Hole, IMH). The normal incidence of this condition is about 0.17%; however, there is a 10-29% chance of development of a macular hole in the fellow eye of patients suffering from unilateral macular hole.

Our hypothesis is that embedded in the topography of the retina is information that can allow for discrimination between healthy eyes and eyes with an increased risk of developing IMH. As such, our work aims to develop a system that allows the automatic identification of these eyes.

DETAILED DESCRIPTION:
A macular hole is a rupture in the macula, the central portion of the retina, responsible for sharp, central vision and hence indispensable for most tasks. In terms of pathogenesis, even though some can be related to trauma, as much as 80% are idiopathic (Idiopathic Macular Hole, IMH). It is theorized that antero-posterior and tangential forces are behind this condition; however, no conclusions have been reached. While the normal incidence of this condition is about 0.17%, there is a 10-29% chance of developing a macular hole in the fellow eye of patients suffering from unilateral macular hole.

Our working hypothesis is that embedded in the topography of the retina is information that can allow for discrimination between healthy eyes and eyes with an increased risk of developing IMH. As such, our study consists on the characterisation of the retinal topography of fellow eyes of patients with unilateral IMH but no other visible retinal pathologies, and of eyes from controls subjects in the same approximate age group. From these topographic maps we acquire a series of features (parameters), and using machine learning techniques create a system that separates eyes into one of the groups - healthy or at risk.

ELIGIBILITY:
Inclusion Criteria:

* normal OCT, with or without vitreous adhesion
* fellow group: unilateral idiopathic macular hole

Exclusion Criteria:

* OCT with vitreous adhesion
* lamellar or pseudoholes
* inner retinal surface alterations
* myopia(>4D)
* glaucoma
* significative media opacity
* previous retina photocoagulation
* any type of intraocular surgery in the last 6 months
* intravitreal medication
* diabetes or neurodegenerative diseases
* macular hole secondary to trauma

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with unilateral idiopathic macular hole and no other visible retinal pathologies.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Macular Topography | at 1 visit
  When a patient that fits into the description of either the case or the control group comes in for a routine visit, a routine optical coherence tomography scan is performed. These scans are non-invasive and common in ophthalmological visits.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Bernardes, Ph.D., Principal Investigator — Institute for Biomedical Imaging and Life Sciences, Faculty of Medicine, University of Coimbra
Locations (7):
- Portugal (7):
  - Braga Hospital, Braga
  - AIBILI - Association for Innovation and Biomedical Research on Light and Image, Coimbra
  - IBILI - Institute for Biomedical Imaging and Life Sciences, Coimbra
  - North Lisbon Hospital Center, Lisbon
  - St. Maria Hospital, Lisbon
  - St. Antonio Hospital, Porto
  - St. Joao Hospital, Porto

REFERENCES:
- [Result] H. Pereira; M. Alfaiate; T. Santos; L. Pedrosa; M. Mendes; R. Venâncio; J. Figueira; R. Bernardes: Identification of Eyes at Risk of Developing Idiopathic Macular Holes by Support Vector Machines. IBILI Meeting 2011, December 2011
- [Result] P. Rodrigues; T. Santos; H. Pereira; J. Figueira; R. Bernardes: Identification of Eyes at Risk of Developing Idiopathic Macular Holes by Support Vector Machines. DOI: 10.1109/ENBENG.2012.6331372
- [Result] J. Figueira; H. Pereira; M. Alfaiate; A. R. Santos; T. Santos; L. Pedrosa; M. Mendes; R. Venâncio; R. Bernardes: Identification of Eyes at Risk of Developing Idiopathic Macular Holes by Support Vector Machines. ARVO Annual Meeting 2012. Invest Ophthalmol Vis Sci 2012;53: E-Abstract 5219.
- [Result] A. S. Silva, T. Santos, S. Simão, J. Figueira, R. Bernardes: Unveiling preclinical idiopathic macular hole formation: structural changes by high-definition OCT and machine learning. V Annual meeting of IBILI, Coimbra, Portugal, December 12-13 2013.
- [Result] Figueira, João; Silva, Ana S. C; Meireles, Angelina; Gomes, Nuno; Ferreira, Natália; Neves, Carlos; Bernardes, Rui. Identificação de Olhos em Risco de Desenvolvimento de Buracos Maculares Idiopáticos (BMI). 56th Congress of the Portuguese Ophthalmology Society. 2013.
- [Result] Silva, Ana S. C; Figueira, João; Simão, Sílvia; Gomes, Nuno; Neves, Carlos; Meireles, Angelina; Ferreira, Natália; Bernardes, Rui. 2014. Unveiling Preclinical Idiopathic Macular Hole Formation Using Support Vector Machines, Proceedings of the Biomedical and Health Informatics International Conference, IEEE - EMB Chapter, 2014.